CLINICAL TRIAL: NCT04150575
Title: A Single-Arm, Open-Label, Multicentre, Phase II Clinical Study to Evaluate Efficacy and Safety of HLX10 (Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection) Combined With Albumin-Bound Paclitaxel in Patients With Advanced Cervical Cancer Who Have Progressive Disease or Intolerable Toxicity After First-Line Standard Chemotherapy
Brief Title: A Clinical Study to Evaluate Efficacy and Safety of HLX10 Combined With Albumin-Bound Paclitaxel in Patients With Advanced Cervical Cancer Who Have Progressive Disease or Intolerable Toxicity After First-Line Standard Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10-011-CC201
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2021-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX10 (Experimental): HLX10+albumin-bound paclitaxel
  Interventions: Drug: HLX10+Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: HLX10+Albumin-Bound Paclitaxel — HLX10: 4.5 mg/kg/3w+Albumin-bound paclitaxel: 260 mg/m2/3w.Albumin-bound paclitaxel may be used for up to 6 cycles, and HLX10 for up to 2 years.
  Other Names: HLX10 is an innovative monoclonal antibody targeting PD-1，developed by Shanghai Henlius Biotech, Inc.

SUMMARY:
This is a single-arm, open-label, multicentre, phase II clinical study.Subjects can only enter this study after they meet the inclusion and exclusion criteria.All enrolled patients will receive the treatment with HLX10 combined with albumin-bound paclitaxel, every 3 weeks, until progressive disease, initiation of new anti-tumour therapy, death, intolerable toxicity. Albumin-bound paclitaxel may be used for up to 6 cycles and HLX10 for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and have signed the informed consent form (ICF);
2. Aged ≥ 18 years and ≤ 75 years at the time of signing the ICF
3. Patients histologically or cytologically diagnosed with cervical cancer (pathology report is required and pathological types are cervical squamous cell carcinoma, adenocarcinoma, and adenosquamous carcinoma).
4. Patients with advanced cervical cancer who have experienced progressive disease or relapse after receiving standard treatment (first-line chemotherapy must be included) or who are intolerant to first-line chemotherapy. First-line chemotherapy includes any of the following:

   1. Platinum-based drugs + taxanes;
   2. Platinum-based drugs + topotecan;
   3. Taxanes + topotecan.
5. The radiological examination during screening confirms the presence of at least one measurable lesion evaluated according to the RECIST v1.1(IRRC).
6. Patients whose tumour specimens are tested positive for PD-L1 expression (CPS ≥ 1).
7. An ECOG score of 0 or 1.
8. Conforming to laboratory measurements;

Exclusion Criteria:

1. Patients who have previously received albumin-bound paclitaxel.
2. Patients with other active malignancies within 5 years or at the same time.
3. Patients who are preparing for or have received an organ or bone marrow transplant.
4. Presence of uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
5. Central nervous system (CNS) or leptomeningeal metastases confirmed by imaging or pathological examination.
6. Class III to IV cardiac insufficiency according to NYHA classification or an LVEF (left ventricular ejection fraction) < 50% by cardiac colour Doppler.

8.With human immunodeficiency virus (HIV) infection. 9.With active pulmonary tuberculosis. 10.Have received any T-cell costimulatory or immune checkpoint therapy, including but not limited to cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors, or other agents that target T cells.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 21 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 2 years
  Objective response rate(assessed by independent radiological review committee (IRRC) based on the RECIST Version 1.1)

SECONDARY OUTCOMES:
ORR | up to 2 years
  Objective response rate (ORR) (assessed by IRRC as per iRECIST, and by the investigator as per RECIST v1.1 and iRECIST, respectively)
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years
  Progression-free survival (PFS) (assessed by IRRC and the investigator as per RECIST v1.1 and iRECIST, respectively)
6-month PFS rate | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 6 months
  6-month progression-free survival rate
OS | from the date of first dose until the date of death from any cause，assessed up to 2 years
  Overall survival
6-month OS rate | from the date of first dose until the date of 6-month
  6-month overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: lingying wu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] An J, Li X, Wang J, Zhu L, An R, Jiang K, Huang Y, Wang K, Li G, Wang C, Yuan J, Hou X, Yang G, Li J, Wang Q, Zhu J, Wu L. Efficacy and safety of serplulimab plus nab-paclitaxel in previously treated patients with PD-L1-positive advanced cervical cancer: a phase II, single-arm study. Front Immunol. 2023 Apr 21;14:1142256. doi: 10.3389/fimmu.2023.1142256. eCollection 2023. PMID 37153587